CLINICAL TRIAL: NCT01520363
Title: Placebo Controlled Trial of Dextromethorphan in Rett Syndrome
Acronym: PCTDMRTT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: The Johns Hopkins Institute for Clinical and Translational Research (ICTR) (Unknown)
Responsible Party: Principal Investigator, SakkuBai Naidu, M.D., Professor of Neurology and Pediatrics, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FD-004247-01
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; RTT; MECP2; dextromethorphan; DM
MeSH Terms: conditions — Rett Syndrome | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study drug-dextromethorphan (DM) (Active Comparator): MECP2 mutation positive subjects randomized to receive DM
  Interventions: Drug: dextromethorphan
- Placebo group (Placebo Comparator): MECP2 positive subjects randomized to the placebo compound
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dextromethorphan — The DM group will take 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study. The pharmacists will dispense the DM to the study participants.
  Other Names: Delsym
  Arms: Study drug-dextromethorphan (DM)
Drug: placebo — The placebo will be dispensed to equal the volume of DM of 5mg/kg/day. It is taken orally in 2 divided doses 12 hours apart during the study period of 3 months. The Research pharmacist will dispense the placebo to the participants.
  Arms: Placebo group

SUMMARY:
Dr. Sakkubai Naidu, Principal Investigator, is initiating a double blinded placebo controlled clinical drug trial using dextromethorphan (DM) in Rett Syndrome (RTT), at the Pediatric Clinical Research Unit (PCRU) of the Johns Hopkins Hospital/Kennedy Krieger Institute. Funding source , FDA-00PD

It has been shown that receptors for a certain brain chemical called glutamate, in particular the NMDA type, are increased in the brain of young RTT patients (<10 years of age). This chemical and its receptors, when in excess, cause harmful over-stimulation of nerve cells in the brain, contributing in part to the seizures, behavioral problems, and learning disabilities in RTT.

The investigators propose to initiate a specific treatment using DM to counter/block the effects of this brain chemical and its excessive receptors to improve the ill effects of increased glutamate/NMDA receptors, because of DM's identified ability to block NMDA receptors. DM is available for human consumption. Infants and children with respiratory infections and cough, as well as non-ketotic hyperglycinemia, are treated with DM, which has been well tolerated.

DETAILED DESCRIPTION:
The study will last for 3 months and will be limited to MECP2 mutation-positive children, one year - 9.99 years of age. This clinical trial, which is a placebo-controlled study, will randomize patients to the drug or placebo to determine the benefits of DM vs placebo on cognition, behavior, or seizures if present.

Your child will stay twice in the Pediatric Clinical Research Unit (PCRU) at Johns Hopkins ICTR, for 3 days during each admission. The first hospital stay will be for 3 days, before she starts the DM or placebo. The follow-up 3-day hospital stay will be 3 months after she starts taking DM or placebo. There will also be two interim follow up evaluations at 2 weeks and 1 month after she starts taking the DM or placebo consisting of a neurological evaluation, EKG, and blood work, which can take place at your local doctor's office or at Johns Hopkins, and will be paid for by this study. Our research nurse or research associate will contact you at least weekly during the first month, and at least monthly thereafter until the end of the 3-month study.

ELIGIBILITY:
Inclusion Criteria:

* males and females who have classic or atypical RTT with a proven mutation in the MECP2 gene;
* subjects must be between one year - 10 years of age.

Exclusion Criteria:

* those without an established mutation in the MECP2 gene;
* those with mutations in the MECP2 gene but who have had brain resection or surgical intervention; for example, tumor, hydrocephalus, severe head trauma; or, an associated severe medical illnesses such as vasculopathies, malignancies, diabetes, thyroid dysfunction, etc;
* those on medications that could interact with DM, e.g. MAO inhibitors, SSRI, sibutramine etc. to avoid a serotonin syndrome; quinidine and drugs metabolized by the CYP450 isoform CYP2D6 (e.g. amiodarone, haloperidol, propafenone, thioridazine);
* those proven to be intermediate or slow metabolizers of DM;
* those with reported adverse reactions to DM;
* those whose pregnancy test is positive;
* those showing poor compliance with any aspect of the study;
* foster children.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sakkubai R Naidu, MD, Principal Investigator — The Kennedy Krieger Institute and Johns Hopkins SOM
Locations (1):
- The Johns Hopkins Institute for Clinical and Translational Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 57 participants were consented. Of these 5 were slow metabolizers who did not meet post consent eligibility criteria.
Period: Overall Study
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group
Started | 26 | 26
Completed | 24 | 26
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 26 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.75 (2.52) | 4.91 (1.91) | 4.83 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
  Canada | 0 | 1 | 1
  Mexico | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Mullen; Visual Reception Sub-scale Scores, Pre- and Post-Intervention
Description: The Mullen Scales of Early Learning (MULLEN) Visual reception subscale raw scores range from Minimum=0 to Maximum=50. A higher score is a better outcome. Age equivalents from 1 month to 70 months can be computed for each subscale separately.
Time Frame: Initial evaluation and at the end of the 3 month trial
Population: Mutation positive participants who are fast metabolizers at baseline. 2 were noncompliant and removed from the study drug group. At 3 months 22 were analyzed in the study drug group and 25 in the placebo group due to incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive DM at baseline
  dextromethorphan: The DM group will take 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study. The pharmacists will dispense the DM to the study participants.
- Placebo Group: MECP2 positive subjects randomized to the placebo at baseline
  placebo: The placebo will be dispensed to equal the volume of DM of 5mg/kg/day. It is taken orally in 2 divided doses 12 hours apart during the study period of 3 months. The Research pharmacist will dispense the placebo to the participants.
- Study Drug Group at 3 Months: MECP2 mutation positive subjects randomized to DM at 3 months
- Placebo at 3 Months: MECP2 mutation positive subjects randomized to placebo at 3 months
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 5.45 (3.419) | 6.61 (6.308) | 6.64 (7.135) | 6.57 (5.008)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = .211, t-test, 2 sided; df=21; Mean Difference (Net) = -1.182, 95% CI 2-sided [-3.086 to .722], Standard Deviation 4.294; t= -1.291; p=.211
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = .949, t-test, 2 sided; df=22; Median Difference (Final Values) = .043, 95% CI 2-sided [-1.345 to 1.432], Standard Error of Mean .670

2. Primary Outcome: Change in Mullen; Fine Motor Sub-scale Scores, Pre- and Post-Intervention
Description: The Mullen Scales of Early Learning (MULLEN) Fine motor scale raw scores range from Minimum=0 to Maximum=49. A higher score is a better outcome. Age equivalents from 1 month to 70 months can be computed for each subscale separately.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 5.38 (5.5) | 7.00 (6.474) | 5.05 (6.103) | 7.04 (6.564)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = .541, t-test, 2 sided — df=20; df=20; Mean Difference (Final Values) = 0.333, 95% CI 2-sided [-0.785 to 1.451], Standard Deviation 2.456; t=0.622; p=.541
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = .946, t-test, 2 sided — df=23; Mean Difference (Net) = -.042, 95% CI 2-sided [-1.290 to 1.206], Standard Deviation 2.956; t=-.069; p=0.946

3. Primary Outcome: Change in Mullen; Receptive Language Subscale Scores, Pre- and Post-Intervention
Description: The Mullen Scales of Early Learning (MULLEN) Receptive Language scale raw scores range from Minimum=0 to Maximum=50. A higher score is a better outcome. Age equivalents from 1 month to 70 months can be computed for each subscale separately.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 6.45 (5.307) | 6.95 (5.269) | 6.68 (5.472) | 6.55 (6.085)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = .736, t-test, 2 sided; df=21; Mean Difference (Net) = -0.227, 95% CI 2-sided [-1.609 to 1.154], Standard Deviation 3.116; t=-0.342; p=0.736
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = .589, t-test, 2 sided; Mean Difference (Net) = 0.409, 95% CI 2-sided [-1.143 to 1.961], Standard Deviation 3.500; t=0.548; p=0.589

4. Primary Outcome: Change in Mullen, Expressive Language Sub-scale Scores, Pre- and Post-Intervention
Description: The Mullen Scales of Early Learning (MULLEN) Expressive Language scale raw scores range from Minimum=0 to Maximum=50. A higher score is a better outcome. Age equivalents from 1 month to 70 months can be computed for each subscale separately.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 5.33 (3.665) | 6.73 (3.8) | 6.76 (5.504) | 7.29 (7.123)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = .05, t-test, 2 sided; df=20; Mean Difference (Net) = -1.429, 95% CI 2-sided [-2.886 to 0.029], Standard Deviation 3.203; t=-2.044; p=0.05
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = 0.958, t-test, 2 sided; Mean Difference (Net) = 0.042, 95% CI 2-sided [-1.589 to 1.672], Standard Deviation 3.862; t=0.053; p=0.958

5. Secondary Outcome: Change in VABS: Motor Skills Domain Scores, Pre- and Post-Intervention
Description: Vineland Adaptive Behavior Scales-II (VABS): Motor Skills Domain Scores individual items are scored on a Likert scale from 2=Usually, 1=Sometimes or Partially, 0= Seldom or Never. Motor Skills Domain raw scores range from: Minimum=0 to Maximum=100. A higher score is a better outcome.
Time Frame: Baseline evaluation and at the end of the 3 month study
Population: MECP2 Mutation positive participants who are fast metabolizers were randomized to placebo or DM at baseline. Two participants in the baseline DM group were noncompliant and removed from the study at baseline. At 3 months 22 were analyzed in the DM study drug group and 25 in the placebo group due to incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) at baseline: The DM group will take 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study.
- Placebo Group: MECP2 positive subjects randomized to the placebo compound at baseline. The placebo will be dispensed to equal the volume of DM of 5mg/kg/day. It is taken orally in 2 divided doses 12 hours apart during the study period of 3 months.
- Study Drug-dextromethorphan (DM) at 3 Months: MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) who completed study assessments at the 3 month time point.
- Placebo Group at 3 Months: MECP2 positive subjects randomized to the placebo compound who completed the assessments at the 3 month time point.
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 9.86 (3.821) | 11.36 (4.838) | 9.64 (3.959) | 11.12 (4.755)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug-dextromethorphan (DM) at 3 Months; Test type: Superiority; p = 0.488, t-test, 2 sided; df=21; Median Difference (Net) = 0.227, 95% CI 2-sided [-0.442 to 0.897], Standard Deviation 1.510; t=0.706; p=0.488
Statistical Analysis 2: Comparison: Placebo Group vs Placebo Group at 3 Months; Test type: Superiority; p = 0.442, t-test, 2 sided; df=24; Median Difference (Net) = 0.24, 95% CI 2-sided [-0.394 to 0.874], Standard Deviation 1.535; t=0.782; p=0.442

6. Secondary Outcome: Change in VABS:Daily Living Skills Domain Scores, Pre- and Post-Intervention
Description: Vineland Adaptive Behavior Scales-II (VABS): Daily Living Skills Domain individual items are scored on a Likert scale from 2=Usually, 1=Sometimes or Partially, 0= Seldom or Never. The Daily Living Skills Domain measures personal behavior as well as domestic and community interaction skills. Daily Living Skills Domain raw scores range from Minimum=0 to Maximum=218.
Time Frame: Baseline and at the end of the 3 month trial
Population: 52 MECP2 Mutation positive participants who are fast metabolizers were enrolled in the study. Two participants in the baseline DM group were noncompliant and removed from the study at baseline. At 3 months 22 were analyzed in the DM study drug group and 25 in the placebo group due to incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) at baseline: The DM group took 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study.
- Placebo Group: MECP2 positive subjects randomized to the placebo compound at baseline: The placebo was dispensed to equal the volume of DM of 5mg/kg/day. It is taken orally in 2 divided doses 12 hours apart during the study period of 3 months. The Research pharmacist dispensed the placebo to the participants.
- Study Drug-dextromethorphan (DM) at 3 Months: MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) who completed the study at 3 months
- Placebo Group at 3 Months: MECP2 positive subjects randomized to the placebo compound were still active in the study at 3 months.
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 21.64 (6.939) | 21.00 (5.307) | 20.95 (6.388) | 19.84 (4.589)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug-dextromethorphan (DM) at 3 Months; Test type: Superiority; p = 0.182, t-test, 2 sided; df=21; Mean Difference (Net) = 0.682, 95% CI 2-sided [-0.346 to 1.709], Standard Deviation 2.317; t=1.380; p=0.182
Statistical Analysis 2: Comparison: Placebo Group vs Placebo Group at 3 Months; Test type: Superiority; p < 0.005, t-test, 2 sided; df=24; Mean Difference (Net) = 1.160, 95% CI 2-sided [0.391 to 1.929], Standard Deviation 1.864; t=3.112; p=0.005

7. Secondary Outcome: Change in VABS: Socialization Domain Scores, Pre- and Post-Intervention
Description: Vineland Adaptive Behavior Scales-II (VABS): Socialization Domain. Critical behaviors are scored on a Likert scale from 2=Usually, 1=Sometimes or Partially, 0= Seldom or Never. Socialization Domain raw scores range from: Minimum=0 to Maximum=152. A higher score is a better outcome.
Time Frame: Baseline and at the end of the 3 month trial
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) at baseline: The DM group will take 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study. The pharmacists dispensed the DM to the study participants.
- Study Drug-dextromethorphan (DM) at 3 Months: MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) at 3 month time period.
- Placebo Group at 3 Months: MECP2 mutation positive subjects randomized to receive DM placebo at 3 month time period.
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 24.14 (5.557) | 22.96 (4.954) | 24.05 (6.514) | 22.48 (5.524)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug-dextromethorphan (DM) at 3 Months; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Net) = .091, 95% CI 2-sided [-1.463 to 1.644], Standard Deviation 3.504; t=0.122; p=0.90
Statistical Analysis 2: Comparison: Placebo Group vs Placebo Group at 3 Months; Test type: Superiority; p = 0.356, t-test, 2 sided; df=24; Mean Difference (Net) = 0.480, 95% CI 2-sided [-0.573 to 1.533], Standard Deviation 2.551; t=0.941; p=0.356

8. Secondary Outcome: Change in VABS:Communication Domain Scores, Pre- and Post-Intervention
Description: Vineland Adaptive Behavior Scales (VABS)-II Communication Domain Scores. The Communication Domain evaluates the receptive, expressive, and written communication skills of the child. Critical behaviors in each Subdomain item are rated as 2=Usually, 1=Sometimes or Partially, 0= Seldom or Never. Communication Domain raw scores range from: Minimum=0 to Maximum=198. A higher score is a better outcome.
Time Frame: Baseline and at the end of the 3 month trial
Population: 52 MECP2 Mutation positive participants who are fast metabolizers were enrolled at baseline. Two participants in the baseline DM group were noncompliant and removed from the study. At 3 months 22 were analyzed in the DM study drug group and 25 in the placebo group due to incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) at baseline: The DM group will take 5mg/kg/day orally in 2 divided doses 12 hours apart for the 3 month period of the study. The pharmacists will dispense the DM to the study participants.
- Study Drug-dextromethorphan (DM) at 3 Months: MECP2 mutation positive subjects randomized to receive DM (dextromethorphan) and active in study at 3 month time point.
- Placebo Group at 3 Months: MECP2 mutation positive subjects randomized to receive Placebo and active in study at 3 month time point.
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 18.05 (4.146) | 18.08 (4.261) | 17.91 (5.032) | 17.96 (4.835)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug-dextromethorphan (DM) at 3 Months; Test type: Superiority; p = 0.836, t-test, 2 sided; Mean Difference (Net) = 0.136, 95% CI 2-sided [-1.220 to 1.493], Standard Deviation 3.060; t=0.209; p=0.836
Statistical Analysis 2: Comparison: Placebo Group vs Placebo Group at 3 Months; Test type: Superiority; p = 0.826, t-test, 2 sided; df=24; Mean Difference (Net) = 0.120, 95% CI 2-sided [-0.993 to 1.233], Standard Deviation 2.698; t=0.222; p=0.826

9. Secondary Outcome: Change in Ghuman-Folstein Screen for Social Interaction (SSI) Score, Pre- and Post-Intervention.
Description: The Ghuman-Folstein Screen for Social Interaction (SSI) assesses the change in behavior and temperament dysregulation as a total score.
  The score ranges from 0-162, with 0 being most Impaired /has the strongest autism features and 162 having no impairment/no autism features.
Time Frame: Initial evaluation and at the end of the 3 month study. The test lasts 45 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 22 | 24 | 22 | 24
units on a scale | 73.1 (22.86) | 71.3 (17.26) | 73.1 (25.97) | 68.0 (16.21)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Placebo Group vs Study Drug Group at 3 Months vs Placebo at 3 Months; Test type: Superiority; p = 0.42, t-test, 2 sided; Mean Difference (Net) = -3.38, 95% CI 2-sided [-11.80 to 5.05], Standard Error of Mean 4.18

10. Secondary Outcome: Change in Rett Syndrome Behavior Questionnaire Score, Pre- and Post-Intervention
Description: The Rett Syndrome Behavior Questionnaire (RSBQ) total score was assessed. The total score ranges from 0 to 90, with 0 exhibiting no Rett syndrome related symptoms and 90 showing the greatest amount of symptoms (worse outcome).
Time Frame: Initial evaluation and at the end of the 3 month study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 22 | 24 | 22 | 24
units on a scale | 33.8 (13.21) | 33.3 (12.26) | 33.8 (13.21) | 33.3 (12.26)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Placebo Group vs Study Drug-dextromethorphan (DM) at 3 Months vs Placebo Group at 3 Months; Test type: Superiority; p < 0.73, t-test, 2 sided; Mean Difference (Net) = -1.03, 95% CI 2-sided [-7.02 to 4.96], Standard Error of Mean 2.97

11. Other Pre Specified Outcome: Change in PedsQL School Functioning Subscale Score, Pre- and Post-Intervention
Description: Pediatric Quality of Life Inventory (PedsQL version 4). School Functioning subscale. 5-point Likert scale from 0 (Never) to 4 (Almost always); Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better Health Related Quality of Life (QOL).
Time Frame: Baseline evaluation and at the end of the 3 month study
Population: MECP2 Mutation positive participants who are fast metabolizers were randomized to placebo or DM at baseline. Two participants in the baseline DM group were noncompliant and removed from the study at baseline. At 3 months, 22 were analyzed in the DM study drug group and 25 in the placebo group due to incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study Drug-dextromethorphan (DM): MECP2 mutation positive subjects randomized to receive dextromethorphan(DM) at baseline
- Placebo Group: MECP2 positive subjects randomized to the placebo at baseline.
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 64.231 (23.3682) | 49.583 (20.3793) | 55.769 (25.2782) | 44.592 (14.2084)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = 0.371, t-test, 2 sided; df=12; Mean Difference (Net) = 8.4615, 95% CI 2-sided [-11.3603 to 28.2834], Standard Deviation 32.8016; t=0.903; p=0.371
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = 0.358, t-test, 2 sided; df=11; Mean Difference (Net) = 4.9917, 95% CI 2-sided [-6.4553 to 16.4387], Standard Deviation 18.0163 — t=0.960; p=0.358

12. Other Pre Specified Outcome: Change in PedsQL Total Score, Pre- and Post-Intervention
Description: Pediatric Quality of Life Inventory (PedsQL version 4) total score. Each item is rated on a 5-point Likert scale from 0 (Never) to 4 (Almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The Total Score is the sum of all the items over the number of items answered on all the Scales. Higher scores indicate better HRQOL.
Time Frame: Baseline evaluation and at the end of the 3 month study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 54.018 (18.5915) | 54.157 (14.9519) | 50.9235 (19.11019) | 51.7286 (18.83983)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = 0.603, t-test, 2 sided; df=16; Mean Difference (Net) = 3.09412, 95% CI 2-sided [-9.27756 to 15.46580], Standard Deviation 24.06228 — t=0.530; p=0.603
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = 0.432, t-test, 2 sided; df=13; Mean Difference (Net) = 2.42857, 95% CI 2-sided [-4.04665 to 8.90380], Standard Deviation 11.21479 — t=0.810; p=0.432

13. Other Pre Specified Outcome: Change in PedsQL Social Functioning Subscale Score, Pre- and Post-Intervention
Description: Pediatric Quality of Life Inventory (PedsQL version 4). Social Functioning subscale. 5-point Likert scale from 0 (Never) to 4 (Almost always); Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better Health Related Quality of Life (QOL).
Time Frame: Baseline and at the end of the 3 month trial
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 58.53 (21.849) | 54.64 (18.341) | 46.76 (16.002) | 47.14 (20.448)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = 0.083, t-test, 2 sided; df=16; Mean Difference (Net) = 11.765, 95% CI 2-sided [-1.745 to 25.275], Standard Deviation 26.276; t=1.846; p=0.083
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = 0.073, t-test, 2 sided; df=13; Mean Difference (Net) = 7.500, 95% CI 2-sided [-0.802 to 15.802], Standard Deviation 14.378; t=1.952; p=0.073

14. Other Pre Specified Outcome: Change in PedsQL Emotional Functioning Subscale Score, Pre- and Post-Intervention
Description: Pediatric Quality of Life Inventory (PedsQL version 4). Emotional Functioning subscale. 5-point Likert scale from 0 (Never) to 4 (Almost always); Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better Health Related Quality of Life (QOL).
Time Frame: Baseline evaluation and at the end of the 3 month study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 72.37 (17.979) | 68.93 (13.182) | 68.621 (24.3816) | 68.214 (113.8129)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug-dextromethorphan (DM) at 3 Months; Test type: Superiority; p = 0.549, t-test, 2 sided; df=18; Mean Difference (Net) = 3.7474, 95% CI 2-sided [-9.1269 to 16.6217], Standard Deviation 26.7110 — t=0.612; p=0.549
Statistical Analysis 2: Comparison: Placebo Group vs Placebo Group at 3 Months; Test type: Superiority; p = 0.874, t-test, 2 sided; df=13; Mean Difference (Net) = 0.7143, 95% CI 2-sided [-8.8174 to 10.2460], Standard Deviation 16.5084 — t=0.162; p=0.874

15. Other Pre Specified Outcome: Change in PedsQL Physical Functioning Subscale Score, Pre- and Post-Intervention
Description: Pediatric Quality of Life Inventory (PedsQL version 4). Physical Functioning subscale. 5-point Likert scale from 0 (Never) to 4 (Almost always); Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better Health Related Quality of Life (QOL).
Time Frame: Initial evaluation and at the end of the 3 month study
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 24 | 26 | 22 | 25
score on a scale | 42.717 (30.3026) | 48.973 (29.5643) | 38.900 (29.7848) | 48.133 (34.9777)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Study Drug Group at 3 Months; Test type: Superiority; p = 0.693, t-test, 2 sided; df=17; Mean Difference (Net) = 3.8167, 95% CI 2-sided [-16.2046 to 23.8379], Standard Deviation 40.2609 — t=0.402; p=0.693
Statistical Analysis 2: Comparison: Placebo Group vs Placebo at 3 Months; Test type: Superiority; p = 0.909, t-test, 2 sided; df=14; Mean Difference (Net) = 0.8400, 95% CI 2-sided [-14.6102 to 16.2902], Standard Deviation 27.8994 — t=0.117; p=0.909

16. Other Pre Specified Outcome: Change in Seizure Frequency, Pre- and Post-Intervention, 0-4 Year Age Group
Description: Change in Frequency of seizure count baseline to follow-up for children aged 0-4 years
Time Frame: Baseline evaluation and at the end of the 3 month study
Population: Children enrolled at baseline aged 0 to 4 years
Measure: Mean (Standard Deviation); unit: seizure count
Groups:
- Study Drug-dextromethorphan (DM) at 3 Months: MECP2 mutation positive subjects randomized to DM at 3 months.
- Placebo Group at 3 Months: MECP2 mutation positive subjects randomized to placebo at 3 months,
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug-dextromethorphan (DM) at 3 Months | Placebo Group at 3 Months
Number analyzed (Participants) | 11 | 10 | 11 | 10
seizure count | 3 (1.41) | 3.2 (1.32) | 3.7 (.90) | 3.1 (1.45)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Placebo Group vs Study Drug-dextromethorphan (DM) at 3 Months vs Placebo Group at 3 Months; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Net) = -0.83, 95% CI 2-sided [-2.17 to 0.52], Standard Error of Mean 0.64

17. Other Pre Specified Outcome: Change in Seizure Frequency, Pre-and Post-Intervention, 5-10 Year Age Group
Description: Change in Frequency of seizures baseline to follow-up for children aged 5-10 years
Time Frame: Baseline evaluation and at the end of the 3 month study
Measure: Mean (Standard Deviation); unit: seizure count
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
Number analyzed (Participants) | 13 | 16 | 11 | 16
seizure count | 3.6 (1.19) | 2.8 (1.47) | 3.36 (1.12) | 3.37 (1.20)
Statistical Analysis 1: Comparison: Study Drug-dextromethorphan (DM) vs Placebo Group vs Study Drug Group at 3 Months vs Placebo at 3 Months; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Net) = 0.74, 95% CI 2-sided [-0.66 to 2.15], Standard Error of Mean 0.68

ADVERSE EVENTS:
Arm/Group | Study Drug-dextromethorphan (DM) | Placebo Group | Study Drug Group at 3 Months | Placebo at 3 Months
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 18/24 | 22/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug-dextromethorphan (DM) (N=26) | Placebo Group (N=26) | Study Drug Group at 3 Months (N=24) | Placebo at 3 Months (N=26)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (8) | 11 (11)
seizures (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Increased alkaline phosphatase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
increased platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT01520363/Prot_SAP_000.pdf